CLINICAL TRIAL: NCT01998711
Title: Memory Group Intervention for Mild Cognitive Impairment: Impact of a Memory Group for Older Adults Reporting Memory Difficulties.
Brief Title: Impact of a Memory Group for Older Adults Reporting Memory Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 156/04
Record Dates: First submitted 2005-09-12; First posted 2013-12-02 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2005-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Alzheimer's disease; Mild cognitive impairment; Memory intervention; Strategy use; Memory group
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory group (Experimental): Memory training
  Interventions: Behavioral: Memory group
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Memory group — Five 1-1.5 hour weekly session of memory training
  Arms: Memory group

SUMMARY:
Aims:

To evaluate the efficacy of a brief intensive intervention for persons with mild cognitive impairment, assisted by family members or friends. To equip persons with mild cognitive impairment with specific skills to prevent memory failures and improve the capacity of patients and families to cope with everyday memory difficulties.

DETAILED DESCRIPTION:
Participants:

The sample will consist of 60 families who have a family member reporting memory loss and who have recently been assessed within the Cognitive Dementia and Memory Service (CDAMS). Participants will include patients and a family member / close friend. The potential patient participants must have received a diagnosis of mild cognitive impairment following a comprehensive clinical assessment. They must also be English speakers, live in the community, have no evidence of significant visual or auditory impairment, and have no history of diagnosed alcohol or drug abuse or major psychological disorder. Potential family / friend participants are expected to be spouses or adult children.

Brief Description:

Patients and their carers will be assigned to either a 'brief intervention group' or a 'no intervention group'. Over 5 1 1/2 -hour weekly sessions, the brief intervention group will be taught a memory skills program which emphasises practical strategies for dealing with everyday memory problems. Interactive group discussion and 'take home' exercises are also included. The no intervention group will serve as a control group, and will receive only their usual care from the the memory clinic. At the completion of the study, the brief intervention will be offered to those in the no intervention group.

All participants will complete questionnaires about knowledge of memory techniques, common memory and behaviour problems and emotional health at pre-intervention, post-intervention and after a 3-month follow-up.

Methods of Data Analysis:

Outcome evaluation will be monitored by neuropsychological assessments of memory performance, and subjective self-reports. A 2 x 3 multivariate analysis of variance (MANOVA) will be used to assess differences on the experimental measures between groups (brief intervention, no intervention) across repeated assessment phases (pre-intervention, post-intervention, 3-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

Participant presents with memory complaint Objective memory impairment on neuropsychological tests Normal general cognitive function Adequate activities of daily living Fails to reach criterion for clinical dementia according to NINCDS-ADRDA guidelines Living in the community Absence of significant visual or auditory impairment English speaker -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Neuropsychological measures of memory and attention
Self-report on memory performance in everyday activities
Self-report on use of memory strategies
Informant report on memory performance in everyday activities
Informant report on use of strategies
Assessment of psychological wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Glynda J Kinsella, PhD, Principal Investigator — Caulfield General Medical Centre - Psychology
Locations (1):
- Caulfield General Medical Centre, Melbourne, Victoria, Australia